CLINICAL TRIAL: NCT04808362
Title: A Phase 1/2 Study to Evaluate the Safety, Pharmacokinetics, and Anti-Tumour Activity of the MYC Inhibitor OMO-103 Administered Intravenously in Patients With Advanced Solid Tumours
Brief Title: Phase 1/2 Study to Evaluate Safety, PK and Efficacy of the MYC-Inhibitor OMO-103 in Solid Tumours
Acronym: MYCure
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Phase 1completed; sponsor decided to change strategy to a combination study
Sponsor: Peptomyc S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMO-103-01
Record Dates: First submitted 2021-03-16; First posted 2021-03-22 (Actual); Results first posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Advanced Solid Tumors; Pancreatic Cancer; CRC
Keywords: MYC-Inhibitor; First in human; solid tumor
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: accelerated titration design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OMO-103 (Experimental): OMO-103 will be administered intravenously as 30 min infusion once weekly
  Interventions: Biological: OMO-103

INTERVENTIONS:
Biological: OMO-103 — OMO-103 will be administered intravenously as 30 min infusion once weekly

SUMMARY:
This study is an open label, two-part, First in Human (FIH) Phase 1/2 dose-finding study designed to determine the safety, tolerability, Pharmacokinetics (PK), Pharmacodynamics (PD) and proof-of-concept (POC) of OMO-103 in patients with advanced solid tumours.

DETAILED DESCRIPTION:
This study is an open label, two-part, FIH Phase 1/2 dose-finding study designed to determine the safety, tolerability, PK, PD and proof-of-concept of OMO-103 in patients with advanced solid tumours.

The study consists of two parts:

• Part 1: Dose escalation in patients with advanced solid tumours, including 5 OMO-103 dose levels.

Approximately 11 to 24 patients in total will be enrolled in Part 1, covering 5 dose levels with the primary objective of determining the safety and tolerability of OMO-103 and defining an appropriate dose for further evaluation in Part 2.

The study will start with an accelerated-titration dose-escalation scheme enrolling one evaluable patient per cohort for the first 2 dose levels followed by a classic 3+3 design.

• Part 2: Dose expansion where at least 3 parallel groups of patients with advanced Non Small Cell Lung Cancer (NSCLC), Triple Negative Breast Cancer (TNBC) and Colorectal Cancer (CRC) will be treated at the recommended Phase 2 dose (RP2D) of OMO-103 to further characterise the safety, tolerability, PK, PD and anti-tumour activity of OMO-103.

Approximately 18 patients will be enrolled in each of the 3 parallel groups of patients (NSCLC, TNBC, CRC) in Part 2.

ELIGIBILITY:
Main Inclusion Criteria:

- Male or female patients, 18 years of age or older who sign the informed consent document, are willing and able to comply with the study protocol and have:

Part 1 (Dose Escalation):

- Histologically or cytologically proven advanced solid tumour for which there is no curative therapy and has progressed on Standard of Care (SOC) treatment or is intolerant to or has no available SOC or SOC unacceptable.

Part 2 (Dose Expansion):

- Histologically or cytologically proven advanced NSCLC whose tumours are KRAS-mutated and where the disease has progressed after a chemotherapy and immunotherapy regimen (at least two prior lines of standard therapy), advanced TNBC where the disease has progressed after having received anthracyclines and taxanes (at least two prior lines of standard therapy) and advanced CRC whose tumours are RAS mutated and where the disease has progressed after at least two prior lines of standard therapy.

Parts 1 and 2:

* Patient must have measurable disease as per RECIST v1.1 criteria
* Tumour biopsy (either from the primary tumour or from metastases) during Screening and during Treatment should be obtained from the patients, if feasible.
* Documented progression on or following the last line of therapy.
* ECOG performance status up to 1.
* Life expectancy of ≥12 weeks.
* Adequate organ function

Main Exclusion Criteria:

Parts 1 and 2:

* Systemic anti-cancer therapy within 4 weeks prior to study entry.
* Radiation therapy within 4 weeks prior to study entry. Localised palliative radiotherapy to non-target lesions is allowed.
* Non-malignant systemic disease including cerebrovascular accident (CVA), unstable angina pectoris, unstable atrial fibrillation, unstable cardiac arrhythmia, myocardial infarction in the last 6 months, New York Heart Association (NYHA) Class III or IV heart failure, coagulation abnormalities and clinically significant pulmonary compromise, particularly a requirement for supplemental oxygen use to maintain adequate oxygenation in the previous 6 months.
* Patients with a history of congenital or acquired immunodeficiency syndrome, or currently receiving immunosuppressive therapy >10 mg prednisolone or equivalent. Patients receiving inhaled or topical corticosteroids are eligible.
* Patients with symptomatic or unstable central nervous system (CNS) primary tumour or metastases and/or carcinomatous meningitis. Patients with documented treated CNS metastases stable for at least 4 weeks may be enrolled at the discretion of the Investigator.
* Patients with need of therapeutic anticoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Garralda, MD, PhD, Principal Investigator — University Hospital Vall d´Hebron; Oncology Department
Locations (3):
- Spain (3):
  - University Hospital Vall d´Hebron, Barcelona
  - Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garralda E, Beaulieu ME, Moreno V, Casacuberta-Serra S, Martinez-Martin S, Foradada L, Alonso G, Masso-Valles D, Lopez-Estevez S, Jauset T, Corral de la Fuente E, Doger B, Hernandez T, Perez-Lopez R, Arques O, Castillo Cano V, Morales J, Whitfield JR, Niewel M, Soucek L, Calvo E. MYC targeting by OMO-103 in solid tumors: a phase 1 trial. Nat Med. 2024 Mar;30(3):762-771. doi: 10.1038/s41591-024-02805-1. Epub 2024 Feb 6. PMID 38321218

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 patients at 3 sites
Period: Overall Study
Arm/Group | OMO-103
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | OMO-103
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] — patients older than 18 years
  years | 61 [32 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Spain | 22

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Safety and Tolerability
Description: Phase 1: Number of patients with a DLT; Number of patients with IRRs, AEs /SAEs according to NCI CTCAE v 5;
Time Frame: DLT period was 3 weeks and AEs were assessed for each patient until progression which was in average 3 months;
Population: safety population
Measure: Number; unit: participants
Arm/Group | OMO-103
Number analyzed (Participants) | 22
participants
  DLT DLT | 1
  TEAEs | 18
  SAEs | 9
  IRRs | 10

2. Secondary Outcome: Phase 1: Elimination Half Life (t1/2)
Description: Phase 1: elimination half life (t1/2) was determined via several timepoints from 0 up to 94 hours after end of infusion
Time Frame: 0, 5, 30, 60 min, 1, 2, 6, 24, 48, 76, 94 hours after end of infusion
Population: Safety population
Measure: Mean (Standard Deviation); unit: hours
Groups:
- OMO-103: OMO-103 will be administered intravenously as 30 min infusion once weekly until progression
Arm/Group | OMO-103
Number analyzed (Participants) | 22
hours | 38 (19)

ADVERSE EVENTS:
Time Frame: AE were collected for each patient from signing informed consent until last follow-up which was in average 3 months but varied a lot from 4 day up to 536 days.
Description: no deviation. CTCAE version 5 was used.
Arm/Group | OMO-103
All-Cause Mortality (participants affected / at risk) | 3/22
Serious Adverse Events (participants affected / at risk) | 9/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OMO-103 (N=22)
Bile Duct Obstruction (Gastrointestinal disorders) | 1 (1) — not related, grade 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) — not related, grade 3
Hydrocephalus (Nervous system disorders) | 1 (1) — not related, grade 3
Abdominal pain (Gastrointestinal disorders) | 1 (1) — not related , grade 2
Epigastralgia (Gastrointestinal disorders) | 1 (1) — not related, grade 2
IRR (General disorders) | 1 (1) — related, grade 3
Worsening anemia (Blood and lymphatic system disorders) | 1 (1) — not related, grade 3
Inguinal Hernia (Gastrointestinal disorders) | 1 (1) — not related, grade 3
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — not related, grade 2
Bowel Obstruction (Gastrointestinal disorders) | 1 (1) — not related, grade 3
Back Pain (Injury, poisoning and procedural complications) | 1 (1) — not related , grade 3
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) — not related, grade 3
Hypoglycemia (Endocrine disorders) | 1 (1) — not related, grade 3
Bacteremia (Infections and infestations) | 1 (1) — not related, grade 2
Respiratory Insufficiency (Respiratory, thoracic and mediastinal disorders) | 1 (1) — not related, grade 3
Malignant disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — not related, grade 5
Back Pain (General disorders) | 1 (1) — not related, grade 3
Pericardial Effusion (Cardiac disorders) | 1 (1) — not related, grade 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OMO-103 (N=22)
Infusion Related Reactions IRR (Injury, poisoning and procedural complications) | 10 (43)
Anemia (Blood and lymphatic system disorders) | 7 (8)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Obstipation (Gastrointestinal disorders) | 1 (2)
Anal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Gastroointestinal Disorder (Gastrointestinal disorders) | 3 (3)
General Disorders (General disorders) | 11 (16)
Hepatobiliary Disorder (Hepatobiliary disorders) | 1 (1)
Infections (Infections and infestations) | 4 (7)
Investigations (Investigations) | 6 (14)
Metabolism (Metabolism and nutrition disorders) | 4 (6)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 10 (20)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Nervous System (Nervous system disorders) | 2 (2)
Scrotal Edema (Reproductive system and breast disorders) | 1 (1)
Respiratory Disorder (Respiratory, thoracic and mediastinal disorders) | 4 (8)
Vascular Disorder (Vascular disorders) | 2 (2)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-09-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT04808362/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT04808362/SAP_001.pdf